CLINICAL TRIAL: NCT02117505
Title: A Single-Dose, Open-Label, Randomized, Crossover Study to Assess the Relative Bioavailability of Two JNJ-54781532 Tablet Formulations Under Fed Conditions in Healthy Adult Subjects
Brief Title: A Crossover Study to Evaluate Relative Bioavailability of Two JNJ-54781532 Tablet Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR104088; 54781532ARA1001
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Biological Availability; JNJ-39220675; Healthy; Phase 1
MeSH Terms: interventions — Akacid-medical-formulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Formulation 2 Then Formulation 1) (Experimental): Single-dose of JNJ-54781532 formulation 2 will be administered as 150 milligram (mg) oral tablet in first treatment period; followed by JNJ-54781532 formulation 1 as 150 mg orally (5*30 mg tablet=150 mg) in second treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Formulation 2; Drug: Formulation 1
- Group 2 (Formulation 1 Then Formulation 2) (Experimental): Single-dose of JNJ-54781532 formulation 1 will be administered as 150 mg oral tablet (5*30 mg tablet=150 mg) in first treatment period; followed by JNJ-54781532 formulation 2 as 150 mg oral tablet in second treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Formulation 2; Drug: Formulation 1

INTERVENTIONS:
Drug: Formulation 2 — Single-dose of JNJ-54781532 formulation 2 will be administered as 150 milligram (mg) oral tablet in one of the treatment periods.
  Other Names: JNJ-54781532 Test
Drug: Formulation 1 — Single-dose of JNJ-54781532 formulation 1 will be administered as 150 milligram (mg) oral tablet (5*30 mg tablet=150 mg) in one of the treatment periods.
  Other Names: JNJ-54781532 Reference

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability (the extent to which a drug or other substance becomes available to the body) of JNJ-54781532 formulation 2 (test) compared with JNJ-54781532 formulation 1 (reference) in healthy participants under fed conditions at a single dose of 150 milligram (mg).

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), 2-treatment, 2-period, 2-sequence crossover (participants may receive different interventions sequentially during the trial), and single-center study of JNJ-54781532. The duration of study will be approximately of 5 weeks per participant. The study consists of 3 parts: Screening (that is, 21 days before study commences on Day 1); Open-label Treatment (consists of 2 single-dose treatments, either JNJ-54781532 formulation 1 [reference] or JNJ-54781532 formulation 2 [test]), in subsequent 2-treatment periods, each separated with washout period of 7 days); and End-of-Study (done upon completion of the 72-hour pharmacokinetic sampling on Day 4 of Period 2, or at the time of early withdrawal). All the eligible participants will be randomly assigned to 1 of the 2 treatment sequences to ensure that they receive both of the following treatments, one in each period. Followed by an overnight fast of at least 10 hours participants will be administered with study treatment 30 minutes after high-fat, high-calorie breakfast. Participants will not be allowed to have food until 4 hours of drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Relative bioavailability of two formulations of JNJ-54781532 (test and reference) will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be either: 1) not of childbearing potential: postmenopausal or surgically sterile at screening 2) of child-bearing potential: Must use highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening, and agree to use highly effective contraception throughout the study period, and for 90 days after final study drug administration. Women, who are not heterosexually active at Screening, must agree to utilize a highly-effective method of birth control if they become heterosexually active during their participation in the study
* Must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day (-)1 of Period 1
* Female participants must agree not to donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration
* If a man who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the Investigator (for example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 90 days after receiving the last dose of study drug
* Participants eligible according to the following tuberculosis (TB) screening criteria: 1) following tuberculosis (TB) screening criteria 2) have no signs or symptoms suggestive of active TB upon medical history and/or physical examination 3) have had no recent close contact with a person with active TB 4. Within 2 months prior to the first administration of study agent, have a negative T-spot or QuantiFERON-TB Gold test result

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection
* Participant had major gastrointestinal (GI) surgery
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center on Day (-) 1 of Period 1
* Participant has an aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than or equal to (>=) the upper limit of normal (ULN)
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 1 year before Screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines) at screening or Day (-) 1 of Period 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (tmax) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The tmax is time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Relative Bioavailability of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  Bioavailability means the extent to which the active ingredient of a drug dosage form becomes available at the site of drug action or in a biological medium believed to reflect accessibility to a site of action. Relative bioavailability of single-dose of two formulations of JNJ-54781532 will be compared in healthy participants under fed conditions.
Time to last quantifiable plasma concentration (tlast) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The tlast is the time to last observed quantifiable plasma concentration.
Area Under the Plasma Concentration Percentage (%) Extrapolation of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The percentage of AUC (0-infinity) that is due to extrapolation from Tlast to infinity (AUC%Extrapolation) is calculated by using the formula AUC_%extrapolation = 100*(AUC [0-infinity] minus (AUC [0-last])/(AUC (0-infinity).
Elimination Half-Life (t [1/2] Lambda) of JNJ-54781532 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Adjusted Coefficient of Determination (R^2 adj) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, and 48 hours (h) post-dose of JNJ-54781532 on Day 1
  The coefficient of determination adjusted for the number of points used in the estimation of Lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium